CLINICAL TRIAL: NCT06658847
Title: A Single Center, Randomized, Evaluator Blinded Clinical Study to Evaluate the Effect of a Topical Retinol on Epigenetic Changes and Expression of Certain Genes in the Skin Using Non-invasive Measurements
Brief Title: A Study to Evaluate the Effect of a Topical Retinol on Epigenetic Changes and Expression of Certain Genes in the Skin Using Non-invasive Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CS2024SK100183
Record Dates: First submitted 2024-10-21; First posted 2024-10-26 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Retinoid; Skin Aging; Epigenomics
Keywords: Retinoid; Skin Aging

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Cell (Experimental): Investigational Night Cream plus auxiliary cleanser and sunscreen
  Interventions: Other: Night Cream Usage
- No Intervention (Active Comparator): Auxiliary cleanser and sunscreen only
  Interventions: Other: No Night Cream Usage

INTERVENTIONS:
Other: Night Cream Usage — Participants will use the provided products only on their face and right upper inner arm. The auxiliary cleanser will be used twice per day (morning and evening). The auxiliary sunscreen will be used 15 minutes prior to sun exposure and reapplied after 80 minutes of sweating or swimming. The investigational night cream will be used daily in the evening/at night.
  Arms: Intervention Cell
Other: No Night Cream Usage — Participants will use the provided products only on their face and right upper inner arm. The auxiliary cleanser will be used twice per day (morning and evening). The auxiliary sunscreen will be used 15 minutes prior to sun exposure and reapplied after 80 minutes of sweating or swimming. No night cream will be used.
  Arms: No Intervention

SUMMARY:
This study is being conducted to confirm whether skin tape stripping methodology can identify changes in gene expression (i.e. whether different genes are turned on to make proteins) in aged skin after use of a retinoid.

DETAILED DESCRIPTION:
This is a randomized study. Participants will be randomly assigned to either the intervention cell and receive a cleanser, a sunscreen serum, and a night cream or the control cell and receive a cleanser and a sunscreen serum to use at home for 10 weeks. Participants will be randomized and receive products at Visit 1 (Screening/Baseline) conducted at Day 0 and return to the clinical site at Day 28 for Visit 2, and at Day 71 for Visit 3.

ELIGIBILITY:
Inclusion Criteria:

1. Has clinically determined moderate photodamage (defined as a score of 4 - 6 on a 0- 9-point scale) on the face at Visit 1.
2. Is able to read, write, speak, and understand English.
3. Generally in good health.
4. Intends to complete the study and is willing and able to follow all study instructions.

Exclusion Criteria:

1. Has known allergies or negative reactions to common topical skincare products, adhesives, latex, or ingredients in the study products.
2. Has clinically active bacterial, fungi, or viral skin infection or has frequent skin infections.
3. Presents with a skin condition that may increase risk to the subject, influence study results, or interfere with study evaluations (e.g. acne, psoriasis, eczema, atopic dermatitis, cutaneous xerosis, erythema, active skin cancer, tattoos, scarring, scratches/broken skin, sunburn, excessive hair growth, or very uneven skin tone) as determined by the principal investigator (PI).
4. Has self-perceived sensitive skin.
5. Is a regular (occasional to daily) smoker of cigarettes or user of electronic cigarettes (vaping pens).
6. Is a regular (occasional or frequent) user of tanning beds and/or self-tanning products.
7. Has had a surgical or aesthetic procedure in the last 3 months that can affect facial wrinkles or facial pigmentation (e.g. botulinum toxin (Botox) injections, chemical peels, laser-based therapies to the face, or face lift surgery).
8. Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti- diabetic medication.
9. Is taking a medication that could mask a negative reaction or influence study results, as determined by the PI.
10. Is self-reported to be breastfeeding, pregnant or planning to become pregnant during the study.
11. Has a history of or a current health/other condition/situation which may put the individual at significant risk, influence the study results, or interfere significantly with the individual's participation in the study.
12. Is currently participating in any other clinical study or has participated in any product-use study within 30 days prior to the study visit.
13. Is an employee/contractor or immediate family member of the PI, study site, or Sponsor.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Skin tape stripping. | Baseline (Day 0), Visit 3 (Day 71)
  The investigator will collect skin samples from subjects through a non-invasive method - tape stripping. The tape strips will be analyzed by extracting DNA collected from the epidermal skin cells then use targeted sequencing using 4M CpG sites to further analyze if certain genes (assessment of UV damage, smoking, and biological age ) are turned on or off from retinol use. Baseline samples will be compared to Day 71 samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Consulting Services, PLLC, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No